CLINICAL TRIAL: NCT02521545
Title: A Single-Dose Study in Healthy Volunteers to Assess the Pharmacokinetic Profile of a New Formulation of BIIB061
Brief Title: Single-Dose Study of a New Formulation of BIIB061
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 231HV103
Record Dates: First submitted 2015-07-16; First posted 2015-08-13 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Multiple Sclerosis
Keywords: Oral Remyelination
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BIIB061 (Experimental): Single oral dose of 30 mg BIIB061 of the new formulation
  Interventions: Drug: BIIB061

INTERVENTIONS:
Drug: BIIB061 — Capsule

SUMMARY:
The primary objective of the study is to assess the pharmacokinetic (PK) profile of BIIB061 in the new oral formulation in the fasted state in healthy male and female volunteers. The secondary objective of this study is to evaluate the safety and tolerability of BIIB061 in the new formulation in this study population.

ELIGIBILITY:
Key Inclusion Criteria:

* Males and postmenopausal (defined as no menses for 12 months and confirmed by follicle-stimulating hormone [FSH] levels determined at screening to be in the postmenopausal range) or surgically sterile females.
* All male subjects must practice effective contraception during the study and be willing and able to continue male contraception for 3 months after the dose of study treatment. All male subjects must also be willing to refrain from sperm donation for at least 3 months after their dose of study treatment.
* Must be in good health and have normal vital signs as determined by the Investigator, based on medical history and screening evaluations.
* Body mass index of 18.0 to 30.0 kg/m2, inclusive.

Key Exclusion Criteria:

* History of or positive test result at screening for human immunodeficiency virus, hepatitis C virus antibody, or hepatitis B virus (defined as positive for hepatitis B surface antigen [HBsAg] or hepatitis B core antibody [HBcAb]).
* Prior exposure to BIIB061.
* History of any clinically significant cardiac, endrocrinologic, hematologic, hepatic, gastric, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, oncologic, or other major disease, as determined by the Investigator.
* Treatment with any prescription medication within 28 days prior to and throughout the duration of the study.
* Use of any over-the-counter products, including herbal or alternative health preparations within the 14 days prior to the study
* Enrollment in any interventional clinical study in which an investigational drug, biologic, device, or approved therapy for investigational use is administered or used within 30 days prior to the study
* Any live or attenuated immunization/vaccination given within 30 days prior to the study or planned to be given during the study.
* Blood donation within 30 days prior to the study
* Surgery within 3 months prior to the study

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2015-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
PK parameter - area under the concentration-time curve from time 0 to infinity (AUCinf) | Day 1-4, 6, 10, 14, 21
PK parameter - AUC from time 0 to time of the last measurable concentration (AUClast) | Day 1-4, 6, 10, 14, 21
PK parameter - maximum observed concentration (Cmax) | Day 1-4, 6, 10, 14, 21

SECONDARY OUTCOMES:
PK parameter - Time to reach maximum observed concentration (Tmax) | Day 1-4, 6, 10, 14, 21
PK parameter - half-life (t1/2) | Day 1-4, 6, 10, 14, 21
Incidence of adverse events (AEs) and serious adverse events (SAEs) | Up to 21 days
Assessment of changes from baseline in Clinical laboratory parameters | Up to 21 days
Assessment of clinically relevant abnormalities in Vital signs | Up to 21 days
Assessment of physical examinations | Up to 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Madison, Wisconsin, United States